CLINICAL TRIAL: NCT04051996
Title: A Randomized, Parallel-arm, Phase 2 Clinical Trial of the Combination of Glasdegib (Pf-04449913) With Two Standard Decitabine Regimens for Older Patients With Poor-risk Acute Myeloid Leukemia Who Are Unfit for or Refuse Intensive Chemotherapy (GLAD-AML)
Brief Title: GLAD-AML - Glasdegib (Pf-04449913) With Two Standard Decitabine Regimens for Older Patients With Poor-risk Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to accrue patients following COVID-19 study pause.
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Amer Zeidan, Associate Professor of Internal Medicine (Hematology), Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000024738
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: ACUTE MYELOID LEUKEMIA
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — glasdegib; Decitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DAC5 (Experimental): Glasdegib will be administered at the starting dose of 100 mg orally once daily and continuously in combination with either DAC5 (decitabine 20 mg/m2 IV on a 5-day schedule) or DAC10 (decitabine 20 mg/m2 IV on a 10-day schedule) as per randomization. Treatment will be administered in 28-day cycles.
  Interventions: Drug: Glasdegib; Drug: Decitabine
- DAC10 (Experimental): Glasdegib will be administered at the starting dose of 100 mg orally once daily and continuously in combination with either DAC5 (decitabine 20 mg/m2 IV on a 5-day schedule) or DAC10 (decitabine 20 mg/m2 IV on a 10-day schedule) as per randomization. Treatment will be administered in 28-day cycles.
  Interventions: Drug: Glasdegib; Drug: Decitabine

INTERVENTIONS:
Drug: Glasdegib — Glasdegib will be administered at the starting dose of 100 mg orally once daily.
Drug: Decitabine — Decitabine will be administered per local label and will be administered by IV infusion at a dose of 20 mg/m2/day for either 5 days or 10 days as determined by randomization. Each cycle will be every 28 days.

SUMMARY:
This multi-center, randomized phase 2 study is designed to evaluate the complete remission (including complete remission with incomplete count recovery) rates of glasdegib in combination with either decitabine on a 5-day or 10-day schedule in patients with newly-diagnosed poor-risk AML who either refuse or are ineligible for intensive therapy.

DETAILED DESCRIPTION:
The primary objective of this multi-center, randomized phase 2 study is to determine the response rates, complete remission (CR) and complete remission with incomplete count recovery (CRi), of glasdegib/DAC5 and glasdegib/DAC10 in patients with newly-diagnosed PrAML.

There are two secondary objectives for this study. The first secondary objective is to evaluate the toxicity and safety profiles of glasdegib/DAC5 and glasdegib/DAC10 in patients with newly-diagnosed PrAML. The other secondary objective is to determine the event-free survival (EFS), relapse-free survival (RFS), overall survival (OS), duration of response, bone marrow mutational clearance, and remission clonality of glasdegib/DAC5 and glasdegib/DAC10 in patients with newly-diagnosed PrAML.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a morphologically-confirmed diagnosis of AML according to WHO 2016 classification with poor-risk disease as defined by the cytogenetic or molecular abnormalities (excluding FLT3-mutated AML).
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
* Adequate Renal Function:

  a. Calculated creatinine clearance (determined by MDRD) ≥50mL/min/1.73m2, or serum creatinine <1.5x upper limit of normal (ULN);
* Adequate Liver Function:

  1. Total serum bilirubin ≤ 2.0 x ULN (unless the bilirubin is principally unconjugated and there is strong suspicion of sub-clinical hemolysis or the patient has documented Gilbert's disease);
  2. Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 3.0 x ULN;
  3. Alkaline phosphatase ≤ 3.0 x ULN.
* Serum or urine pregnancy test (for female patients of childbearing potential) with a minimum sensitivity of 25 IU/L or equivalent units of human chorionic gonadotropin (HCG) negative at screening.
* Males and female patients both of childbearing potential and at risk for pregnancy must agree to use two highly effective method(s) of contraception throughout the study and for 180 days after the last dose of decitabine and the last dose of glasdegib, whichever occurs later.
* Female patients who are not of childbearing potential (i.e. meet at least 1 of the following criteria):

  1. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  2. Have medically confirmed ovarian failure;
  3. Have achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal women.

Exclusion Criteria:

* Patients who are candidates for and willing to receive intensive induction chemotherapy.
* Prior use of a hypomethylating agent.
* Prior use of cytotoxic chemotherapy for any myeloid malignancy (prior immunosuppressive therapy is permitted provided that treatment is stopped within 8 weeks from study entry; hydroxyurea is allowed through the end of cycle 1 on study).
* Previous hematopoietic stem cell transplant.
* Prior treatment with a licensed or experimental smoothened inhibitor (SMOi) and/or hypomethylating agent (HMA).
* Participation in a clinical study involving an investigational drug(s) (Phases 1-4) within 4 weeks prior to study entry or within 5 half-lives of the investigational agent, whichever is greater.
* Major surgery or radiation within 12 weeks prior to study entry.
* Patients known to be refractory to platelet or packed red cell transfusions as per institutional guidelines, or who are known to refuse or who are likely to refuse blood product support.
* Treatment with hematopoietic growth factors including: erythropoietin, granulocyte colony stimulating factor (G-CSF), and granulocyte macrophage colony stimulating factor (GM-CSF), or thrombopoietin receptor agonists within 3 weeks prior to study entry.
* Any ongoing medical condition requiring chronic use of moderate to high dose steroids (defined as ≥10 mg/day of prednisone or equipotent dose of another corticosteroid).
* Any anti-cancer treatment within 2 weeks prior to study entry (including hydroxyurea as above).
* Current use or anticipated requirement for drugs that are known moderate to strong CYP3A4 inducers (Appendix 2).
* Presence of concurrent active malignancy requiring active systemic therapy
* Patients with known active, uncontrolled bacterial, fungal or viral infection, including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS) related illness.
* Known uncontrolled central nervous system (CNS) involvement.
* Poorly-controlled active medical conditions that as per investigator judgement would interfere with the conduct of the study.
* Active cardiac dysrhythmias of NCI CTCAE Grade ≥2 (e.g. atrial fibrillation) or QTcF interval >470 msec.
* Pregnant or breastfeeding female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amer M Zeidan, MBBS, Principal Investigator — Yale University - MEDCCC Hematology-Section
Locations (1):
- Yale Cancer Center/Smilow, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DAC5 | DAC10
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 patient was enrolled in the study prior to termination and therefore would be identified through presenting these characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | DAC5 | DAC10 | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: CR/CRi
Description: The complete remission (CR) and complete remission with incomplete count recovery (CRi) combined rate will be defined by the 2017 European LeukemiaNet (ELN) AML response criteria.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | DAC5 | DAC10
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: OS
Description: Overall survival (OS) is defined as the time from date of first study treatment to date of death due to any cause.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | DAC5 | DAC10
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: EFS
Description: Event-free survival (EFS) will be monitored up to 2 years.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | DAC5 | DAC10
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: RFS
Description: Relapse-free survival (RFS) will be monitored up to 2 years.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | DAC5 | DAC10
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to CR/CRi
Description: The time to complete remission (CR) and complete remission with incomplete count recovery (CRi) will be collected as a secondary outcome.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | DAC5 | DAC10
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of CR/CRi
Description: The duration of complete remission (CR) and complete remission with incomplete count recovery (CRi) will be collected as a secondary outcome.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | DAC5 | DAC10
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Bone Marrow Mutational Clearance
Description: Bone marrow mutational clearance of frequently-mutated genes in AML (e.g. NPM1, CEBPA, DNMT3A, RUNX1, TET2, IDH1/2) via next-generation DNA sequencing will be monitored up to 2 years.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | DAC5 | DAC10
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: There was only 1 patient enrolled in the study before termination and therefore there was only 1 treatment arm utilized.
Arm/Group | DAC5 | DAC10
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAC5 (N=1) | DAC10 (N=0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT04051996/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT04051996/ICF_001.pdf